CLINICAL TRIAL: NCT00599638
Title: A TWO WEEK DOUBLE-BLIND PLACEBO-CONTROLLED CROSSOVER STUDY TO COMPARE THE EFFICACY AND SAFETY OF A PREGABALIN/PF-00489791 COMBINATION VERSUS PREGABALIN ALONE IN PATIENTS WITH POST-HERPETIC NEURALGIA
Brief Title: A Study To Compare Pregabalin/PF-00489791 Combination Versus Pregabalin Alone In Post-Herpetic Neuralgia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: B0261002
Record Dates: First submitted 2008-01-04; First posted 2008-01-24 (Estimated); Results first posted 2021-08-05 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-08

CONDITIONS: Postherpetic Neuralgia
MeSH Terms: conditions — Neuralgia, Postherpetic | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (3):
- 1 (Active Comparator)
  Interventions: Drug: pregabalin
- 2 (Experimental)
  Interventions: Drug: pregabalin/PF-00489791
- 3 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: pregabalin — 75mg bid titrating to 150mg bid on day 4
  Arms: 1
Drug: pregabalin/PF-00489791 — Pregabalin 75mg bid titrating to 150mg bid on day 4; PF-00489791: 4mg od titrating to 10mg od on day 4
  Arms: 2
Drug: Placebo — Placebo
  Arms: 3

SUMMARY:
Pregabalin is an alpha-2 delta ligand approved for the treatment of neuropathic pain, however, not all patients will respond to this drug. This study will compare the efficacy of pregabalin when administered with an experimental drug PF-00489791, in patients with post-herpetic neuralgia. The efficacy of this combination will be compared to pregabalin alone.

ELIGIBILITY:
Inclusion Criteria:

* Male or female of non-childbearing potential
* Pain present for more than 3 months after healing of herpes zoster skin rash
* VAS score of >=40mm at screening and baseline visits

Exclusion Criteria:

* Patients with pain conditions which might impair the assessment of postherpetic neuralgia
* Skin conditions in the affected dermatome that could alter sensation other than postherpetic neuralgia
* History or diagnosis of DSM IV major depressive disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2008-04-09 (Actual); Primary Completion 2008-12-16 (Actual); Study Completion 2008-12-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (39):
- United States (39):
  - North Alabama RadioPharmacy, Huntsville, Alabama
  - Tennessee Valley Pain Consultants, Huntsville, Alabama
  - River Region Research, LLC, Tallassee, Alabama
  - Radiant Research, Chandler, Arizona
  - Novara Clinical Research, Mesa, Arizona
  - Community Medical Providers, Clovis, California
  - Sierra Medical Research (Administrative only site), Fresno, California
  - Prime-Care Clinical Research, Mission Viejo, California
  - Parkinson's Disease and Movement Disorders Center of Boca Raton, Boca Raton, Florida
  - Bradenton Research Center, Bradenton, Florida
  - Arthritis Associates of South Florida, Delray Beach, Florida
  - Delray Research Associates, Delray Beach, Florida
  - Office of Laszlo J Mate, M.D., West Palm Beach, Florida
  - American Medical Research, Inc., Oak Brook, Illinois
  - Beacon Clinical Research, Brockton, Massachusetts
  - ICPS Group, Norwood, Massachusetts
  - Neurological Research Center at Hattiesburg Clinic, Hattiesburg, Mississippi
  - CRC of Jackson, Jackson, Mississippi
  - Physician's Surgery Center, Jackson, Mississippi
  - Clinvest, Springfield, Missouri
  - Centennial Park Medical Building, North Platte, Nebraska
  - Neurology Associates of Great Plains, North Platte, Nebraska
  - Finger Lakes Clinical Research, Rochester, New York
  - North State Clinical Research, PLLC, Lenoir, North Carolina
  - The Center for Clinical Research, Winston-Salem, North Carolina
  - Legacy Pharma Research, Bismarck, North Dakota
  - Patient Priority Clinical Sites, LLC, Cincinnati, Ohio
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Mark A. Fisher, MD-Private Practice, Oklahoma City, Oklahoma
  - Absolute Primary Care, P.C., Cranberry Twp., Pennsylvania
  - John P. Murtha Neuroscience and Pain Institute, Johnstown, Pennsylvania
  - Memorial Medical Center, Johnstown, Pennsylvania
  - New England Center for Clinical Research, Cranston, Rhode Island
  - Medical Clinic of North Texas, Arlington, Texas
  - FutureSearch Trials of Neurology, Austin, Texas
  - Futuresearch Trials, Austin, Texas
  - Pinnacle Pain Medicine, Dallas, Texas
  - The Medical Group Of Texas, Fort Worth, Texas
  - Medical and Surgical Clinic of Irving, Irving, Texas

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

RESULTS

PARTICIPANT FLOW:
Groups:
- Pregabalin Then Placebo: Participants received 75 milligram (mg) capsule of Pregabalin orally twice daily from Day 1 to Day 3 and 150 mg capsule of Pregabalin orally twice daily from Day 4 to Day 14 in first intervention period followed by placebo matched to Pregabalin twice daily from Day 1 to Day 14 in second intervention period. A washout period of at least 14 days was maintained between each intervention period. Participants had follow up of 1 week.
- Placebo Then Pregabalin: Participants received placebo matched to Pregabalin twice daily from Day 1 to Day 14 in first intervention period followed by Pregabalin 75 mg capsule orally twice daily from Day 1 to Day 3 and 150 mg capsule of Pregabalin orally twice daily from Day 4 to Day 14 in second intervention period. A washout period of at least 14 days was maintained between each intervention period. Participants had follow up of 1 week.
- Pregabalin + Placebo Then Pregabalin + PF-00489791: Participants received 75 mg capsule of Pregabalin orally twice daily from Day 1 to Day 3 and 150 mg capsule of Pregabalin orally twice daily from Day 4 to Day 14 along with placebo matched to PF-00489791 orally once daily from Day 1 to Day 14 in first intervention period. In second intervention period participants received 75 mg capsule of Pregabalin orally twice daily from Day 1 to Day 3 and 150 mg capsule of Pregabalin orally twice daily from Day 4 to Day 14 along with two tablets of 2 mg PF-00489791 orally once daily from Day 1 to Day 3 and 10 mg tablet of PF-00489791 orally once daily from Day 4 to Day 14. A washout period of at least 14 days was maintained between each intervention period. Participants had follow up of 1 week.
- Pregabalin + PF-00489791 Then Pregabalin + Placebo: Participants received 75 mg capsule of Pregabalin orally twice daily from Day 1 to Day 3 and 150 mg capsule of Pregabalin orally twice daily from Day 4 to Day 14 along with two tablets of 2 mg PF-00489791 orally once daily from Day 1 to Day 3 and 10 mg tablet of PF-00489791 orally once daily from Day 4 to Day 14 in first intervention period. In second intervention period participants received 75 mg capsule of Pregabalin orally twice daily from Day 1 to Day 3 and 150 mg capsule of Pregabalin orally twice daily from Day 4 to Day 14 along with a placebo matched to PF-00489791 orally once daily from Day 1 to Day 14. A washout period of at least 14 days was maintained between each intervention period. Participants had follow up of 1 week.
Period: First Intervention Period (2 Weeks)
Arm/Group | Pregabalin Then Placebo | Placebo Then Pregabalin | Pregabalin + Placebo Then Pregabalin + PF-00489791 | Pregabalin + PF-00489791 Then Pregabalin + Placebo
Started | 16 | 14 | 20 | 22
Treated | 16 | 13 | 20 | 21
Completed | 14 | 12 | 17 | 17
Not Completed | 2 | 2 | 3 | 5
Not completed — Adverse Event | 1 | 0 | 3 | 2
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 1 | 0 | 1
Not completed — Randomized but not Treated | 0 | 1 | 0 | 1
Period: Washout Period (2 Weeks)
Arm/Group | Pregabalin Then Placebo | Placebo Then Pregabalin | Pregabalin + Placebo Then Pregabalin + PF-00489791 | Pregabalin + PF-00489791 Then Pregabalin + Placebo
Started | 14 | 12 | 17 | 17
Completed | 13 | 11 | 17 | 14
Not Completed | 1 | 1 | 0 | 3
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 1 | 0 | 0
Period: Second Intervention Period (2 Weeks)
Arm/Group | Pregabalin Then Placebo | Placebo Then Pregabalin | Pregabalin + Placebo Then Pregabalin + PF-00489791 | Pregabalin + PF-00489791 Then Pregabalin + Placebo
Started | 13 | 11 | 17 | 14
Completed | 12 | 11 | 17 | 14
Not Completed | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who were randomized and had received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pregabalin Then Placebo | Placebo Then Pregabalin | Pregabalin + Placebo Then Pregabalin + PF-00489791 | Pregabalin + PF-00489791 Then Pregabalin + Placebo | Total
Number analyzed (Participants) | 16 | 13 | 20 | 21 | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 8 | 5 | 7 | 27
  >=65 years | 9 | 5 | 15 | 14 | 43
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 13 | 14 | 43
  Male | 8 | 5 | 7 | 7 | 27

OUTCOME MEASURES:

1. Primary Outcome: Mean Pain Score on Daily Pain Rating Scale (DPRS)
Description: Pain was assessed by using a daily pain rating scale that consisted of an 11-point numeric scale ranging from 0 ("no pain") to 10 ("worst possible pain"), higher scores indicate more pain intensity. Participants described their pain during the past 24 hours by choosing the appropriate number between 0 and 10. Self-assessment was performed daily. The mean pain score was defined as the mean of the last 7 daily pain ratings scale scores while taking study medication, at end of each treatment period: Period 1 (Week 2) and Period 2 (Week 6), respectively. Mean pain score had a score range of 0 (no pain) to 10 (worst possible pain), higher scores indicate more pain. Cumulative data of mean pain scores at end of treatment for both the periods was calculated and reported in terms of adjusted mean and standard error.
Time Frame: End of treatment period (included both Week 2 and Week 6)
Population: Full analysis set included all participants who were randomized and had received at least 1 dose of study drug, regardless of whether they had efficacy data and did not have any significant protocol violation. Here, "Overall Number of Participants Analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Pregabalin + PF-00489791: Participants received 75 mg capsule of Pregabalin orally twice daily from Day 1 to Day 3 and 150 mg capsule of Pregabalin orally twice daily from Day 4 to Day 14 along with two tablets of 2 mg PF-00489791 once daily from Day 1 to Day 3 and 10 mg tablet of PF-00489791 once daily from Day 4 to Day 14 in first or second intervention period.
- Pregabalin: Participants received 75 mg capsule of Pregabalin orally twice daily from Day 1 to Day 3 and 150 mg capsule of Pregabalin orally twice daily from Day 4 to Day 14 in first or second intervention period.
- Placebo: Participants received placebo matched to Pregabalin capsule from Day 1 to Day 14 in first or second intervention period.
Arm/Group | Pregabalin + PF-00489791 | Pregabalin | Placebo
Number analyzed (Participants) | 38 | 59 | 25
units on a scale | 4.32 (0.343) | 4.22 (0.253) | 5.57 (0.451)
Statistical Analysis 1: Comparison: Pregabalin + PF-00489791 vs Pregabalin; Test type: Superiority or Other; p = 0.3910, Mixed Models Analysis; Adjusted Mean Difference = 0.08, 80% CI 2-sided [-0.31 to 0.48], Standard Error of Mean 0.306
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis; Adjusted Mean Difference = -1.32, 80% CI 2-sided [-1.78 to -0.86], Standard Error of Mean 0.357

2. Secondary Outcome: Percentage of Participants With Patient Global Impression of Change (PGIC) Score
Description: The PGIC is a participant-rated instrument that measures change in the participants' overall status on a 7-point scale. Scores range from 1 (very much improved) to 7 (very much worse), lower scores indicated more improvement. PGIC was evaluated using 3 categories: improvement (scores 1-3), no change (score 4), and worsening (scores 5-7). In this outcome measure percentage of participants with categories: improved, no change and worsening, based on PGIC score were reported. Cumulative data at end of treatment for both the periods (Period 1 [Week 2] and Period 2 [Week6]) was calculated and reported.
Time Frame: End of treatment period (included both Week 2 and Week 6)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Pregabalin + PF-00489791 | Pregabalin | Placebo
Number analyzed (Participants) | 31 | 54 | 23
percentage of participants
  Improved | 77.42 | 77.78 | 39.13
  No Change | 16.13 | 18.52 | 43.48
  Worse | 6.45 | 3.70 | 17.39
Statistical Analysis 1: Comparison: Pregabalin + PF-00489791 vs Pregabalin; The statistical analysis was performed compositely for all categories; Test type: Superiority or Other; p = 0.4959, Regression, Logistic; Odds Ratio (OR) = 1.0055, 80% CI 2-sided [0.30 to 1.71]
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; The statistical analysis was performed compositely for all categories; Test type: Superiority or Other; p = 0.0011, Regression, Logistic; Odds Ratio (OR) = 5.0763, 80% CI 2-sided [1.69 to 8.46]

3. Secondary Outcome: Pain Visual Analogue Scale (VAS) at Baseline and Week 4
Description: Participants marked intensity of the pain on a scale, ranging from 0 millimeters (mm) = no pain to 100 mm = worst possible pain, where higher scores indicate more pain.
Time Frame: Baseline, Week 4
Population: Full analysis set included all participants who were randomized and had received at least 1 dose of study drug, regardless of whether they had efficacy data and did not have any significant protocol violation. Here, "Number Analyzed" signifies the number of participants who were evaluable at specified time points for each arm, respectively.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Pregabalin + PF-00489791 | Pregabalin | Placebo
Number analyzed (Participants) | 38 | 60 | 25
mm
  Baseline: number analyzed (Participants) | 21 | 36 | 12
  Baseline | 66.48 (10.64) | 65.92 (14.32) | 67.92 (16.37)
  Week 4: number analyzed (Participants) | 17 | 24 | 13
  Week 4 | 60.88 (22.42) | 63.79 (14.33) | 55.92 (22.22)

4. Secondary Outcome: Neuropathic Pain Symptom Inventory (NPSI)
Description: Participant rated 10-item questionnaire to evaluate different symptoms of neuropathic pain (spontaneous pain like [item 1 to 3]: burning, squeezing, pressure; painful attack like [item 4 to 5]: electric shock, stabbing; pain provoked on [item 6 to 8]: light touching, pressure, contact with something cold; abnormal sensations like [item 9 to 10]: pins and needles, tingling). Each item was rated on an 11-point numerical scale range: 0 (absence of pain) to 10 (maximum intensity of pain). Total NPSI scale ranged from 0 (no pain) to 100 (maximum pain). Higher scores indicate a greater intensity of pain. Cumulative data of NPSI scale at end of treatment for both the periods (Period 1 [Week 2] and Period 2 [Week 6]) was calculated and reported in terms of adjusted mean and standard error.
Time Frame: End of treatment period (included both Week 2 and Week 6)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin + PF-00489791 | Pregabalin | Placebo
Number analyzed (Participants) | 35 | 55 | 24
units on a scale | 25.71 (3.134) | 25.87 (2.168) | 35.25 (5.148)
Statistical Analysis 1: Comparison: Pregabalin + PF-00489791 vs Pregabalin; Test type: Superiority or Other; p = 0.3380, Mixed Models Analysis; Adjusted Mean Difference = 1.18, 80% CI 2-sided [-2.47 to 4.84], Standard Error of Mean 2.819
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Test type: Superiority or Other; p = 0.0022, Mixed Models Analysis; Adjusted Mean Difference = -9.65, 80% CI 2-sided [-13.89 to -5.42], Standard Error of Mean 3.268

5. Secondary Outcome: Number of Participants With Clinically Significant Vital Signs Abnormalities
Description: Vital signs abnormalities included sitting, standing: systolic, diastolic blood pressure and heart rate. Clinical significance was judged by investigator.
Time Frame: Baseline up to Week 7
Population: Safety analysis set included all participants who were randomized and had received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Pregabalin + PF-00489791 | Pregabalin | Placebo
Number analyzed (Participants) | 38 | 61 | 26
Participants | 0 | 2 | 1

6. Secondary Outcome: Number of Participants With Clinically Significant Electrocardiogram (ECG) Abnormalities
Description: Criteria for ECG abnormalities: Maximum QTc (corrected QT) interval, QTcB (Bazett's correction formula) and QTcF (Fridericia's correction formula): 450 to less than (<) 480 milliseconds (msec), 480 to <500 msec and greater than equal to (>=) 500 msec; Maximum QTc interval increase from baseline: >=30 to <60 and >=60 (msec); PR interval: >=300 msec and percent change >=25 or 50 percent; QRS complex: percent change >=25 or 50 percent. Clinical significance was judged by investigator.
Time Frame: Baseline up to Week 7
Population: Safety analysis set included all participants who were randomized and had received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Pregabalin + PF-00489791 | Pregabalin | Placebo
Number analyzed (Participants) | 38 | 61 | 26
Participants | 1 | 0 | 0

7. Secondary Outcome: Number of Participants With Clinically Significant Laboratory Abnormalities: Hematology
Description: Criteria for hematology abnormalities included Hemoglobin: <0.8*lower limit of normal (LLN) and hematocrit: <0.8*LLN. Clinical significance was judged by investigator.
Time Frame: Baseline up to Week 7
Population: Safety analysis set included all participants who were randomized and had received at least 1 dose of study medication. Here "Overall Number of Participants Analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Pregabalin + PF-00489791 | Pregabalin | Placebo
Number analyzed (Participants) | 37 | 60 | 26
Participants | 0 | 0 | 0

8. Secondary Outcome: Number of Participants With Clinically Significant Laboratory Abnormalities: Clinical Chemistry
Description: Criteria for clinical chemistry abnormalities included total bilirubin: greater than (>) 1.5*upper limit of normal (ULN); aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase: >3.0*ULN; total protein, albumin: <0.8*LLN or >1.2*ULN; blood urea nitrogen, creatinine: >1.3*ULN; uric acid: >1.2*ULN; sodium: <0.95*LLN or >1.05*ULN; potassium, chloride, calcium: <0.9*LLN or >1.1*ULN; creatine kinase: >2.0*ULN. Clinical significance was judged by investigator.
Time Frame: Baseline up to Week 7
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Pregabalin + PF-00489791 | Pregabalin | Placebo
Number analyzed (Participants) | 37 | 60 | 26
Participants | 0 | 0 | 0

9. Secondary Outcome: Number of Participants With Clinically Significant Laboratory Abnormalities: Urinalysis
Description: Urinalysis abnormalities criteria included: urine specific gravity: <1.003 to >1.030; urine pH: <4.5 to >8; urine glucose, urine ketones, urine proteins, urine blood/hemoglobin: >=1. Clinical significance was judged by investigator.
Time Frame: Baseline up to Week 7
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Pregabalin + PF-00489791 | Pregabalin | Placebo
Number analyzed (Participants) | 37 | 60 | 26
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant or one participant may have experienced both a serious and non-serious event during the study. Safety data was summarized using randomized patients that took at least 1 dose of study medication.
Arm/Group | Pregabalin + PF-00489791 | Pregabalin | Placebo
Serious Adverse Events (participants affected / at risk) | 1/38 | 0/61 | 0/26
Other Adverse Events (participants affected / at risk) | 22/38 | 35/61 | 7/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin + PF-00489791 (N=38) | Pregabalin (N=61) | Placebo (N=26)
Chest discomfort (General disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Pregabalin + PF-00489791 (N=38) | Pregabalin (N=61) | Placebo (N=26)
Blood disorder (Blood and lymphatic system disorders) | 1 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 1
Lacrimation increased (Eye disorders) | 1 | 1 | 0
Vision blurred (Eye disorders) | 2 | 2 | 0
Visual impairment (Eye disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 4 | 1
Dry mouth (Gastrointestinal disorders) | 2 | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 0
Faecal incontinence (Gastrointestinal disorders) | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 0 | 0
Lip blister (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 1 | 1
Drug withdrawal syndrome (General disorders) | 0 | 1 | 0
Chest pain (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 0 | 5 | 0
Gait disturbance (General disorders) | 0 | 1 | 0
Oedema (General disorders) | 1 | 0 | 0
Oedema peripheral (General disorders) | 2 | 2 | 0
Pain (General disorders) | 0 | 1 | 0
Seasonal allergy (Immune system disorders) | 1 | 0 | 0
Anorectal infection (Infections and infestations) | 0 | 1 | 1
Laryngitis (Infections and infestations) | 0 | 1 | 0
Tooth abscess (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 0
Viral infection (Infections and infestations) | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Blood pressure decreased (Investigations) | 0 | 0 | 1
Blood pressure increased (Investigations) | 2 | 2 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 0 | 0
Weight increased (Investigations) | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Increased appetite (Metabolism and nutrition disorders) | 1 | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 3 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0
Aphasia (Nervous system disorders) | 0 | 3 | 0
Balance disorder (Nervous system disorders) | 2 | 1 | 0
Burning sensation (Nervous system disorders) | 0 | 1 | 0
Disturbance in attention (Nervous system disorders) | 2 | 1 | 0
Dizziness (Nervous system disorders) | 7 | 9 | 0
Dizziness postural (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 3 | 4 | 2
Hyperaesthesia (Nervous system disorders) | 0 | 1 | 0
Lethargy (Nervous system disorders) | 0 | 2 | 0
Memory impairment (Nervous system disorders) | 1 | 1 | 0
Mental impairment (Nervous system disorders) | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0
Sciatica (Nervous system disorders) | 0 | 1 | 0
Somnolence (Nervous system disorders) | 2 | 6 | 0
Speech disorder (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0
Agitation (Psychiatric disorders) | 0 | 1 | 1
Anxiety (Psychiatric disorders) | 1 | 2 | 0
Disorientation (Psychiatric disorders) | 0 | 2 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0
Libido decreased (Psychiatric disorders) | 0 | 1 | 0
Nervousness (Psychiatric disorders) | 0 | 1 | 0
Withdrawal syndrome (Psychiatric disorders) | 0 | 1 | 0
Hypertonic bladder (Renal and urinary disorders) | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0
Nocturia (Renal and urinary disorders) | 0 | 1 | 0
Penis disorder (Reproductive system and breast disorders) | 0/14 | 1/27 | 1/13 — This event was gender specific.
Testicular pain (Reproductive system and breast disorders) | 0/14 | 1/27 | 0/13 — This event was gender specific.
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Sinus operation (Surgical and medical procedures) | 1 | 0 | 0
Flushing (Vascular disorders) | 1 | 0 | 0
Hot flush (Vascular disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.